CLINICAL TRIAL: NCT02275130
Title: Assessment of the Functional Effect of Treatment of Glottic Insufficiency With Injection Technique With the Use of Calcium Hydroxyapatite
Brief Title: Functional Effect of Treatment of Glottic Insufficiency With Calcium Hydroxyapatite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FNO-ENT-Radiesse Voice; DRO-FNOs/2014 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2014-10-15; First posted 2014-10-27 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Glottic Insufficiency
Keywords: glottic insufficiency; calcium hydroxyapatite; augmentation of vocal cords with injection technique
MeSH Terms: interventions — Durapatite; Prolaryn Plus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium Hydroxyapatite (Experimental): 30 patients with glottic insufficiency treated operatively with augmentation of vocal cords with injection technique
  Interventions: Procedure: Calcium Hydroxyapatite; Device: Radiesse Voice (Calcium Hydroxyapatite)

INTERVENTIONS:
Procedure: Calcium Hydroxyapatite — Surgical augmentation of the vocal cords with injection of calcium hydroxyapatite
  Other Names: Radiesse Voice
Device: Radiesse Voice (Calcium Hydroxyapatite)

SUMMARY:
The voice is an indispensable source of human communication. Current time puts high demands on the quality of voice in most professions. Organic or functional changes of vocal cords associated with their insufficiency lead to a deterioration of voice quality, voice fatigue, hoarseness or breathing difficulties. This has adverse psychological, social and economic consequences for the patient, the employer and its surroundings. The injection techniques can be performed under general and local anaesthesia. The defined injectable substance is inserted directly in the vocal cords, which increases its volume and results in an almost immediate improvement of the voice quality. For injection can be used various materials, e.g. autologous fat, calcium hydroxyapatite, silicone, and others. Injection techniques are less invasive, associated with less perioperative morbidity. Operation can be also performed under local anaesthesia in selected patients, therefore is preferred for patients with multiple comorbidities and risk of general anaesthesia.

DETAILED DESCRIPTION:
The causes of glottic insufficiency (vocal fold insufficiency) may be paresis (immobility) of one or both vocal folds (of iatrogenic aetiology after thyroid surgery, neck operations or ingrowth of malignant tumours of the chest or mediastinum, idiopathic after viral infections or central neuropathy) and atrophy (loss of mass) of the vocal cords, which particularly affect older patients. Surgical treatment of insufficiency is indicated for patients in whom conservative treatment is ineffective.

Surgical treatment of vocal fold insufficiency is carried out in two ways:

* By thyroplasty type I, operations performed mostly under general anaesthesia, by the external access to the neck with the insertion of a silicone block through the thyroid cartilage into the space next to the vocal cords, which moves it medially.
* Augmentation of the vocal cords, at which an insertion of an own (fat, cartilage, etc.) or a foreign (Gore-Tex, silicone, etc.) material laterally from the vocal cords can facilitate a change in the position of the vocal cords. In recent years, more and more so-called augmentation injection techniques are preferred.

While thyroplasty has been carried out in the Czech Republic for 10-15 years, the clinicians have had only limited experience with the injection techniques, which has been used for several years only and information about the functional results are still insufficient to date.

The working hypotheses

* Augmentation of vocal folds with hydroxyapatite leads to significant improvements in subjective and objective parameters of voice
* Augmentation of vocal folds with hydroxyapatite is a method comparable with other methods of treatment of glottic insufficiency (thyroplasty type 1, vocal folds augmentation with autologous fat)
* Augmentation of vocal folds with hydroxyapatite can be performed under local anaesthesia The objective of the study is to determine the functional effect of augmented vocal folds with calcium hydroxyapatite ("Radiesse Voice") by comparing selected defined parameters preoperatively and postoperatively.

Other anticipated benefits of the study treatment include improving the quality of life of patients (improved voice quality, breathing, improve of mental state, preventing of social isolation and economic consequences). It will also lead to the introduction of new processes, materials and methods. It is also possible to expect shortening of the hospital stay, decrease in postoperative morbidity, and the possibility to perform the procedure on an outpatient basis.

The study has been designed as a prospective study, which is in conformity with the principles and guidelines of the Helsinki Declaration, good clinical practice and has been approved by the Ethical Committee of the University Hospital Ostrava.

The patients enrolled in the study will be followed for the period of twelve months.

Timetable of the study procedures and controls:

Preoperative examination:

* Demographic data on age, sex, weight, height, smoking, cause of insufficiency
* Questionnaires Voice Handicap Index (VHI)
* Stroboscopy examination (assessment of the size of insufficiency)
* Voice Analysis (Vospector Program - Breathable, Hoarseness, total grade of dysphonia, Maximum Phonation time, Dysphonia Severity Index - based on examination of the voice range

Examination 3 months postoperatively

* Questionnaires Voice Handicap Index (VHI)
* High-speed laryngoscopy, stroboscopy and videokymography (assessment of the size of insufficiency)
* Voice Analysis (Vospector Program - Breathable, Hoarseness, total grade of dysphonia, Maximum Phonation time, Dysphonia Severity Index - based on examination of the voice range

Examination 6 months after surgery

* Questionnaires Voice Handicap Index (VHI)
* High-speed laryngoscopy, stroboscopy and videokymography (assessment of the size of insufficiency)
* Voice Analysis (Vospector Program - Breathable, Hoarseness, total grade of dysphonia, Maximum Phonation time, Dysphonia Severity Index - based on examination of the voice range.

Examination 12 months after surgery (optional examination with cooperative patients)

* Questionnaires Voice Handicap Index (VHI)
* High-speed laryngoscopy, stroboscopy and videokymography (assessment of the size of insufficiency)
* Voice Analysis (Vospector Program - Breathable, Hoarseness, total grade of dysphonia, Maximum Phonation time, Dysphonia Severity Index - based on examination of the voice range.

Statistical data processing For statistical evaluation descriptive statistics will be used (arithmetical average, standard deflection, frequency tables), X2 test, Fisher's exact test, analysis of variance (ANOVA), calculating of the OR (odds ratio) with 95 % confidence intervals, and logistic regression. Statistical tests will be evaluated at the significance level of 5%. Statistical analysis will be performed in the "Stata 10" programme. Program MS Excel will be used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Insufficiency caused by paresis or atrophy
* Duration of insufficiency of at least six months
* Size of the insufficiency not exceeding three millimetres
* Signing of the informed consent

Exclusion Criteria:

* Size of the insufficiency exceeding three millimetres

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Objective improvement of voice parameters | 32 months
  irregularity, noise, overall severity, jitter, shimmer, GNE

SECONDARY OUTCOMES:
Endoscopic assessment | 32 months
  The presence or absence of insufficiency (YES/NO) will be assessed prior to the surgical intervention and after the intervention, by the means of endoscopy examination

CONTACTS AND LOCATIONS:
Overall Officials: Radana Walderová, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Czech Republic, Czechia